CLINICAL TRIAL: NCT01809444
Title: The Effect of Prednisone Versus Doxycycline in Active, Moderately Severe Graves' Orbitopathy: A Randomized, Multi-center, Double-blind, Parallel-controlled Trial
Brief Title: Prednisone Versus Doxycycline in the Treatment of Graves' Orbitopathy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dan Liang, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5010-doxy
Record Dates: First submitted 2012-12-02; First posted 2013-03-12 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Thyroid Associated Opthalmopathies
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Prednisone; sulfadiazine, tetroxoprim drug combination; Chlortetracycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisone+placebo of Doxycycline (Active Comparator): Prednisone: 50 mg/d for 14 day, tailed by 40 mg/d for 14 day, 30 mg/d for 28 day, 20 mg/d for 28 day, 15 mg/d for 14 day, 10 mg/d for 14 day, in total 16 weeks; Placebo of doxycycline: administered for 16 weeks.
  Interventions: Drug: Prednisone+placebo of Doxycycline
- Doxycycline+placebo of Prednisone (Experimental): Doxycycline: 50 mg/d for 12 weeks, and placebo for another 4 weeks; Placebo of prednisone: administered for 16 weeks.
  Interventions: Drug: Doxycycline+placebo of Prednisone

INTERVENTIONS:
Drug: Prednisone+placebo of Doxycycline — Prednisone: 50 mg/d for 14 day, tailed by 40 mg/d for 14 day, 30 mg/d for 28 day, 20 mg/d for 28 day, 15 mg/d for 14 day, 10 mg/d for 14 day, in total 16 weeks; Placebo of doxycycline: administered for 16 weeks
  Other Names: deltacortisone
  Arms: Prednisone+placebo of Doxycycline
Drug: Doxycycline+placebo of Prednisone — Doxycycline: 50 mg PO per day for 12 weeks, and placebo for another 4 weeks; Placebo of prednisone: administered for 16 weeks.
  Other Names: Dolotard; Tibirox; Biomycin
  Arms: Doxycycline+placebo of Prednisone

SUMMARY:
The aim of this study is to compare the efficacy and safety of prednisone versus sub-antimicrobial dose doxycycline (50 mg/d) in the treatment of active moderate-severe Graves' Orbitopathy (GO).

DETAILED DESCRIPTION:
Graves' orbitopathy is an autoimmune disease characterized by an inflammatory phase followed by fibrosis. Surgery to correct eyelid swelling, proptosis, and diplopia is effective, but can not be done until the inflammatory phase has passed. To arrest the inflammatory phase, several types of immunosuppressive treatments have been investigated. Corticosteroids are the first-choice immunosuppressive treatment, having a successful outcome of 50-70% in patients. However, long time usage of corticosteroids often cause severe side-effects.

Sub-antimicrobial dose doxycycline posses known anti-inflammatory effects that are separate from their antibacterial mode of action. This mode of action has lead to the routine use of sub-antimicrobial dose doxycycline for treating inflammatory or autoimmune diseases, such as rosacea, periodontitis and multiple sclerosis. The mechanism is by inhibiting lymphocyte proliferation and production of colony-stimulating factor, inflammatory cytokines, and immunoglobulins, factors thought to play a role in the orbital autoimmune process. These mechanisms make them, in theory, an attractive option of doxycycline for treating Graves' Orbitopathy. In addition, only few adverse events were reported when doxycycline were administered for 3 months in patients with periodontitis or rosacea.

We propose to compare the effect and safety of sub-antimicrobial dose doxycycline versus prednisone for treating non-sight threatening, moderate-severe, inflammatory GO.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Graves' Orbitopathy (as defined by Bartley and Gorman)

  * Eyelid retraction (upper eyelid margin at or above the superior corneoscleral limbus in primary gaze without frontalis muscle contraction) in association with any one of the following:

    * Thyroid dysfunction or abnormal regulation (increased serum thyroxine or triiodothyronine level, decreased serum thyroid stimulating hormone level, absence of thyroid radioiodine uptake suppression after administration of triiodothyronine, or the presence of thyroid stimulating immunoglobulins in serum)
    * Exophthalmos
    * Extraocular muscle involvement (restrictive myopathy or objective evidence of enlarged muscles)
    * Optic nerve dysfunction (abnormal visual acuity, color vision, pupillary reaction or perimetry not attributable to other causes) OR
  * Thyroid dysfunction or abnormal regulation in association with any one of the following:

    * Exophthalmos
    * Extraocular muscle involvement
    * Optic nerve dysfunction
* Moderate-severe GO According to EUGOGO statement, patients with moderate-severe GO usually have any one or more of the following：lid retraction≥2mm, moderate or severe soft tissue involvement, exophthalmos≥3mm above normal for race and gender, inconstant, or constant diplopia.
* Clinical activity score ≥ 3
* Being euthyroid for at least 1 months before the date of inclusion
* Must be able to swallow tablets
* Written informed consent is obtained

Exclusion Criteria:

* Mild Graves' Orbitopathy
* Sight-threatening Graves' Orbitopathy
* Clinical activity score < 3
* Previous treatment for GO Oral steroids, intravenous steroids, radiotherapy
* Pregnant females as determined by positive (serum or urine) human chorionic gonadotrophin (hCG) test at screening or prior to dosing, or lactating females
* Uncontrolled diabetes or hypertension
* History of mental / psychiatric disorder
* Hepatic dysfunction (Albumin (Alb) , Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) and Alkaline phosphates levels must be within normal range for eligibility)
* Renal impairment (Urea and Creatinine levels must be within normal range)
* Doxycycline or Prednisone allergy or intolerance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Estimated)
Dates: Start 2012-11; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Overall treatment response | 24 weeks
  Overall treatment response was graded as: improvement, deterioration, and no success.
  1. Improvement, when at least one major criteria or two minor criteria were achieved, in absence of deterioration of any criterion in that observed eye.Three major criteria were: improvement in diplopia grade (disappearance or change in grade); improvement of ≥8 degrees in any direction of eye movements; reduction of three points or more in CAS. Four minor criteria were: reduction of 2 mm or more in eyelid aperture; reduction of 2 mm or more in proptosis; improvement in grade of soft tissue swelling; decrease in CAS by at least two points.
  2. Deterioration, defined as occurrence of DON, and/or worsening of soft tissue swelling, and/or worsening of diplopia, and/or an increase of ≥2 mm in lid aperture, and/or an increase of ≥2 mm in proptosis, and/or a decrease of ≥8 degrees in duction.
  3. No success was defined if there was no change or the changes did not reach the improvement criteria.

SECONDARY OUTCOMES:
• Health related quality of life questionnaires (GO-QoL) | 24 weeks
• Safety and tolerability as assessed by adverse events, vital signs | 48 weeks
• Quantitative changes of rectus diameter measured by MRI scan | 24 weeks
Relapse | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dan Liang, MD, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, China; Liya Wang, MD, Principal Investigator — Henan Eye Institue, Henan, China; Luosheng Tang, MD, Principal Investigator — The second xiangya hospital of central south university, Hunan, China
Locations (6):
- China (6):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Zhongshan Ophthalmic Center, Guangzhou, Guangdong
  - JOINT SHANTOU INTERNATIONALL EYE CENTER of Shantou University and the Chinese University of Hong Kong, Shantou, Guangdong
  - Shenzhen Eye Hospital, Shenzhen, Guangdong
  - Henan Eye Institue, Henan, China, Zhengzhou, Henan
  - The second xiangya hospital of central south university, Changsha, Hunan

REFERENCES:
- See also: Genetics Home Reference related topics: Lenz microphthalmia syndrome oculofacioc — http://ghr.nlm.nih.gov/
- See also: MedlinePlus related topics: Antibiotics Eye Diseases Thyroid Diseases — http://www.nlm.nih.gov/medlineplus
- See also: U.S. FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks